CLINICAL TRIAL: NCT00694174
Title: Skin Blood Flow Changes Using Laser Doppler Imager for Assessment of Pain and Analgesia in Newborn Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Michigan (Other)
Responsible Party: Victoria Tutag Lehr, Pharm.D., Children's Hospital of Michigan, The Detroit Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 027505MP4F
Record Dates: First submitted 2008-06-04; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Procedural Pain
Keywords: Procedural Pain in Newborn Infants; newborn infant; acute procedural pain; skin blood flow changes; sucrose analgesia; laser doppler imager; neonatal infant pain scale
MeSH Terms: conditions — Pain, Procedural | interventions — Sucrose; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 2 ml sucrose 25% oral solution one time only dose by mouth
  Interventions: Drug: sucrose 24% oral solution
- 2 (Placebo Comparator): sterile water 2 ml one time only dose given by mouth prior to heel lance
  Interventions: Drug: sterile water

INTERVENTIONS:
Drug: sucrose 24% oral solution — sucrose 24% oral solution 2 ml one time only dose administered by mouth prior to heel lance
  Other Names: Oral sucrose solution
  Arms: 1
Drug: sterile water — sterile water 2 ml single dose to be administered orally one time prior to heel lance
  Other Names: sterile water U.S.P.
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether an instrument, the Laser Doppler Imager, is able to measure the effect of pain related changes in skin blood flow in newborn infants. The study will also determine whether the use of sucrose (sugar water) when given by mouth has any effect on pain related skin blood flow changes.

DETAILED DESCRIPTION:
During the last 25 years evidence that newborns can experience pain has been increasing. Painful procedures (injections, heel lances, and circumcisions) are part of normal routine newborn care. Studies have demonstrated that newborns have increased sensitivity to pain when compared with older children and adults. Pain assessment and management is an important component in the overall care of the newborn infant and safe, effective analgesics are needed.

Pain assessment is complicated by the infants' verbal and cognitive limitations. Heart rate, blood pressure and oxygen saturation are commonly monitored in the nursery in response to pain, yet these parameters are affected by handling, illness, medications, as well as by pain. Skin blood flow has been documented to increase in premature newborns undergoing painful procedures in the Newborn Intensive Care Nursery. In the present study, Laser Doppler Imager technology will be used to define changes in skin blood flow response to heel lance and oral sucrose administration in normal newborn infants.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from parent or legal guardian.
* Term, newborn infant, between 1 and 7 days of age.
* Appropriate for gestational age (weight 5th through 95th percentile).

Exclusion Criteria:

* Small or large for gestational age (weight<5th or >95th percentile).
* Physical or biochemical abnormalities.
* History of maternal drug dependence.
* Apgar score <7 at 5 minutes.
* Current use of analgesics.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
skin blood flow response (perfusion units, PU) | immediately prior to heel lance, at heel lance, 5 minutes post heel lance (3 time points)

SECONDARY OUTCOMES:
Heart rate | 10 minutes prior to heel lance, immediately prior to heel lance, at heel lance, 5 minutes post end heel lance
Blood pressure | 10 minutes prior to heel lance, 5 minutes after heel lance
Respiratory rate | 10 minutes prior to heel lance, immediatel prior to heel lance, at time of heel lance, 5 minutes post end heel lance
axillary temperature | 10 minutes prior to heel lance, immediately prior to heel lance, at time of heel lance, 5 minutes post end heel lance
oxygen saturation (SaO2) | 10 minutes prior to heel lance, immediately prior to heel lance, at time of heel lance, 5 minutes post end heel lance
Neonatal Infant Pain Score | 10 minutes prior to heel lance, immediately prior to heel lance, at time of heel lance, 5 minutes post end heel lance

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Tutag Lehr, Pharm.D., Principal Investigator — Children's Hospital of Michigan, The Detroit Medical Center, Wayne State University; Josef Cortez, M.D., Principal Investigator — Hutzel Women's University Hospital, The Detroit Medical Center, Wayne State University
Locations (1):
- Hutzel Women's University Hospital, The Detroit Medical Center, Detroit, Michigan, United States

REFERENCES:
- [Background] Martin H, Lindblad B, Norman M. Endothelial function in newborn infants is related to folate levels and birth weight. Pediatrics. 2007 Jun;119(6):1152-8. doi: 10.1542/peds.2006-2706. PMID 17545383
- [Background] Holland AJ, Martin HC, Cass DT. Laser Doppler imaging prediction of burn wound outcome in children. Burns. 2002 Feb;28(1):11-7. doi: 10.1016/s0305-4179(01)00064-x. PMID 11834324
- [Background] Johnston CC, Stevens BJ. Experience in a neonatal intensive care unit affects pain response. Pediatrics. 1996 Nov;98(5):925-30. PMID 8909487
- [Background] Gonsalves S, Mercer J. Physiological correlates of painful stimulation in preterm infants. Clin J Pain. 1993 Jun;9(2):88-93. doi: 10.1097/00002508-199306000-00003. PMID 8358144
- [Background] Moustogiannis AN, Raju TN, Roohey T, McCulloch KM. Intravenous morphine attenuates pain induced changes in skin blood flow in newborn infants. Neurol Res. 1996 Oct;18(5):440-4. doi: 10.1080/01616412.1996.11740448. PMID 8916058
- [Background] McCulloch KM, Ji SA, Raju TN. Skin blood flow changes during routine nursery procedures. Early Hum Dev. 1995 Apr 14;41(2):147-56. doi: 10.1016/0378-3782(95)01617-c. PMID 7601018
- [Background] Bonamy AK, Martin H, Jorneskog G, Norman M. Lower skin capillary density, normal endothelial function and higher blood pressure in children born preterm. J Intern Med. 2007 Dec;262(6):635-42. doi: 10.1111/j.1365-2796.2007.01868.x. Epub 2007 Nov 7. PMID 17986202
- [Background] Anand KJ, Johnston CC, Oberlander TF, Taddio A, Lehr VT, Walco GA. Analgesia and local anesthesia during invasive procedures in the neonate. Clin Ther. 2005 Jun;27(6):844-76. doi: 10.1016/j.clinthera.2005.06.018. PMID 16117989
- [Background] Anand KJ, Aranda JV, Berde CB, Buckman S, Capparelli EV, Carlo W, Hummel P, Johnston CC, Lantos J, Tutag-Lehr V, Lynn AM, Maxwell LG, Oberlander TF, Raju TN, Soriano SG, Taddio A, Walco GA. Summary proceedings from the neonatal pain-control group. Pediatrics. 2006 Mar;117(3 Pt 2):S9-S22. doi: 10.1542/peds.2005-0620C. PMID 16777824
- [Derived] Tutag Lehr V, Cortez J, Grever W, Cepeda E, Thomas R, Aranda JV. Randomized placebo-controlled trial of sucrose analgesia on neonatal skin blood flow and pain response during heel lance. Clin J Pain. 2015 May;31(5):451-8. doi: 10.1097/AJP.0000000000000126. PMID 24918475